CLINICAL TRIAL: NCT02994030
Title: Biomarker for Duchenne Muscular Dystrophy: An International, Multicenter, Observational, Longitudinal Protocol
Brief Title: Biomarker for Duchenne Muscular Dystrophy
Acronym: BioDuchenne
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BDMD 6-2018
Record Dates: First submitted 2016-11-22; First posted 2016-12-15 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Increased Lordosis/Scoliosis; Hyporeflexia; Duchenne Muscular Dystrophy; Red-Green Color Blindness; Lordosis; Scoliosis; Muscular Atrophy; Muscular Weakness
Keywords: Duchenne Disease; Biomarker
MeSH Terms: conditions — Scoliosis; Reflex, Abnormal; Muscular Dystrophy, Duchenne; Color Vision Defects; Lordosis; Muscular Atrophy; Muscle Weakness; Tabes Dorsalis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Duchenne Muscular Dystrophy (DMD): Participants diagnosed with Duchenne Muscular Dystrophy (DMD) aged between 2 months and 50 years

SUMMARY:
International, multicenter, observational, longitudinal study to identify biomarker/s for Duchenne Muscular Dystropy (DMD) and to explore the clinical robustness, specificity, and long-term variability of these biomarker/s.

DETAILED DESCRIPTION:
Duchenne Muscular Dystrophy (DMD) is a devastating inherited neuromuscular disorder that affects 1 in 3300 live male births (females can be mildly affected carriers). DMD causes progressive weakness and loss of muscle mass, with symptoms usually appearing in early childhood. DMD arises from mutations in the DMD gene that codes for dystrophin.

The DMD gene is located on the short arm of chromosome X (locus Xp21) and codes for dystrophin, containing 3685 amino acid residues. 60-65% of DMD mutations are large dele-tions, 10-30% are nonsense and frame-shift mutations, 5-15% are duplications, and 2% are intronic or 5'- and 3'-UTR alterations.Dystrophin aggregates as a homotetramer in the skeletal muscles or associates with actin and Dystrophin-Associated Glycoproteins (DAGs), forming a stable complex that interacts with laminin in the extracellular matrix. Dystrophin is considered a key structural element in the muscle fiber, whose primary function is to stabilize plasma mem-brane, while the DAGs maintain the sarcolemmal stability by mediating the complex interactions of the muscle membrane and extracellular environment. The low levels of dystrophin lead to cellular instability and progressive leakage of intracellular components, explaining the characteristically high levels of creatine phosphokinase (CPK) in the blood of DMD patients.

Biomarkers serve as measurable indicators of normal biological or pathological processes. They are typically directly linked to genetic variants in specific genes and can predict, diagnose, monitor, and assess the severity of a disease. It is the goal of this study to identify, validate, and monitor biochemical markers from DMD affected participants.

ELIGIBILITY:
INCLUSION CRITERIA

* Informed consent is obtained from the parent/ legal guardian
* The participant is aged between 2 months and 50 years
* The diagnosis of DMD is genetically confirmed by CENTOGENE

EXCLUSION CRITERIA

* Informed consent is not obtained from the parent/ legal guardian.
* The participant is younger than 2 months or older than 50 years
* The diagnosis of DMD is not genetically confirmed by CENTOGENE

Ages: 2 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with Duchenne Muscular Dystrophy (DMD)
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Identification of DMD biomarker/s | 36 weeks
  All samples will be analyzed for the identification of biomarker/s via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

SECONDARY OUTCOMES:
Exploring the clinical robustness, specificity, and long-term variability of DMD biomarker/s | 36 months
  Samples will be analyzed for the identified biomarker candidates via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof.Dr, Study Chair — Centogene GmbH
Locations (12):
- University Hospital Center Mother Teresa, Tirana, Albania
- Egypt (5):
  - Department of Pediatric,Faculty of Medicine, Alexandria University Children's Hospital, Alexandria
  - Ain Shams University-Medical Genetics, Cairo
  - Ain Shams University, Cairo
  - Ain Shams Univirsity, Cairo
  - Departmnet of Pediatrics, Tanta University, Tanta
- Departmnet of Molecular and Medical Genetics, Tbilisi State Medical University, Tbilisi, Georgia
- Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala, India
- American of science and technology, Beirut, Lebanon
- Department of Pediatric Gastroenterology and Hepatology, The Children's Hospital and Institute of Child Health, Lahore, Pakistan
- Emergency Hospital for Children "Louis Turcanu", Timișoara, Romania
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided